CLINICAL TRIAL: NCT02569359
Title: Efficacy and Safety of Shea Nut Oil in Hemophilic Arthropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: participants were not recruited enough
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tsung-Ying Li, Attending Physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-104-05-041
Record Dates: First submitted 2015-10-01; First posted 2015-10-06 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia; Hemophilic Arthropathy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shea nut oil (Experimental): 100% shea nut oil extract with 75% triterpene esters. Daily dosage is three 750 mg soft gel capsules (2250 mg/per day) taken in the morning for 3 months
  Interventions: Dietary Supplement: shea nut oil extract
- Placebo (Placebo Comparator): placebo which comprised 100% canola oil or starch mixed soybean oil
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: shea nut oil extract
  Arms: Shea nut oil
Other: Placebo
  Arms: Placebo

SUMMARY:
Recurrent hemarthrosis results in synovitis and destructive arthropathy in hemophilic patients. Prophylactic replacement, physical therapy, cyclooxygenase-2 (COX-2) inhibitors, corticosteroids, and radionucleotide synovectomy are some of the typical modalities used in the managements hemophilic synovitis and arthropathy. In clinical practice, the choice of non-steroidal anti-inflammatory drugs (NSAIDs) also needs to take into consideration the risk for cardiovascular events and should be used at the lowest effective dose and for the shortest duration.This study will investigate the safety and efficacy of Shea nut oil for the treatment of hemophilic arthropathy.

DETAILED DESCRIPTION:
Hemophilia is an X-linked recessive bleeding disorder caused by a deficiency of coagulation factor VIII (hemophilia A) or IX (hemophilia B). Severe hemophilia patients may have frequent spontaneous bleeding episodes such as joint and muscle bleeding. Repeated joint bleeding leads to chronic synovitis, cartilage damage and bony destruction, which is associated with range of motion (ROM) limitation, pain, muscle atrophy, functional impairment and poor quality of life. Around 80% of all spontaneous joint bleeds occur in the ankles, knees and elbows. Hemophilic arthropathy is a multifactorial event and there is evidence to suggest that iron may play a major role with release of cytokines such as Interleukin-1, Interleukin-6, and tumor necrosis factor-α (TNF-α) eading to chronic proliferative synovitis, hypervascularity, and progressive arthropathy . Prophylactic replacement , physical therapy, COX-2 inhibitors , corticosteroids, and radionucleotide synovectomy are some of the typical modalities used in the managements hemophilic synovitis and arthropathy. The onset of joint bleedings in severe hemophilia occurs approximately 23 months of age and arthropathy could be marked in adolescents or young adults. Some hemophilia patients may either not be good candidates for surgery or may prefer not to have surgery. The traditional Africans have used African Shea tree and shea nuts oil extracts to treat arthritis. Shea nut oil contains are a mixture of fatty acid and cinnamic acid esters of such triterpene alcohols as α-amyrine, β-amyrine, butyrospermol, lupeol and to aminor extent, sterols, aliphatic alcohols, and karitene. Triterpene alcohols such as lupeol and α/β-amyrine have been shown to possess anti-inflammatory effects, especially in their esterified forms. In 1998, US Food and Drug Administration approved shea nut oil as a safe food additive. The shea nut oil used in this trial is a patented concentrate containing approximately 50% triterpenes derived from the seed of the shea tree, Vitellaria paradoxa. The most abundant triterpenes in shea nut oil areα-amyrin(54.6%), β-amyrin(12.3%), Lupeol(17%) plus their dihydro-derivatives. Cheras et al. reported that shea nut oil extract treatment over the 15 weeks of their random double-blind study in upper quartile of 89 osteoarthritis patients was effective in decreasing inflammation marker TNF-α (23.9% vs 6%, treatment vs placebo) and cartilage degradation marker C-terminal crosslinked telopeptide type II collagen (CTX-II) (28.7% vs an increase of 17.6%, treatment vs placebo). Chen and his colleagues carried out a 16-week study in 33 patients with osteoarthritis of knee joint and found shea nut oil was effective in increasing activity and thickness of vastus medialis, and decreasing pain and stiffness of knee joint. Late stage of hemophilic arthropathy is characterized by advanced cartilage degeneration and joint destruction. These effects on cartilage and subchondral bone are degenerative and inflammatory in nature, similar to the changes in osteoarthritis. Management of chronic hemophilic arthropathy is difficult. NSAIDs have been used with caution in patients with bleeding disorders because of their inhibition of platelet function and gastrointestinal side effects. In clinical practice, the choice of NSAIDs also needs to take into consideration the risk for cardiovascular events and should be used at the lowest effective dose and for the shortest duration. This study will investigate the safety and efficacy of Shea nut oil for the treatment of hemophilic arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* age 20 years and above
* hemophilia A or B patients who reported painful (VAS ≥ 3) hemophilic arthropathy in ankles, elbows or knees for at least 6 months.

Exclusion Criteria:

* presence of joint infections
* any surgery on the joint in preceding 6 months
* intra-articular HA injection within the past 6 months
* history of rheumatoid arthritis,
* gouty arthropathy
* presence of neoplasm,
* allergy to shea nut oil production
* use of corticosteroids within 3 weeks prior to baseline and throughout the study
* use of anti-inflammatory agents 3 weeks prior to baseline and for the duration of the study,
* history of trauma associated with the signal joint,
* liver function tests greater than twice the upper limit of normal at baseline
* history of alcohol or substance abuse.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Pain (visual analogue scale) and Change from Baseline Pain at 1 &3 months | baseline, 1 month, 3 months
  The pain intensity will be evaluated subjectively on a visual analogue scale (0-100mm).

SECONDARY OUTCOMES:
CTX-II (ng/mmol creatinine) and Change from Baseline at 1 & 3 months | baseline, 1 month, 3 months
  C-telopeptide fragments of type II collagen (CTX-II) in urine is a measure of type II collagen degradation and a biological marker of arthropathy.
Tumor Necrosis Factor alpha (pg/mL) and Change from Baseline at 1 & 3 months | baseline, 1 month, 3 months
  TNF-alpha are one of inflammatory mediators that increase following hemarthrosis in hemophilic mice. Plasma samples will tested by ELISA.
Ultrasonographic synovial thickness (mm) and Change from Baseline at 1 &3 months | baseline, 1 month, 3 months
  Synovial thickness (mm) by ultrasonography were evaluated from the lateral, middle, and medial aspects of the anterior suprapatellar recess
Synovial hyperemia (score) and Change from Baseline at 1& 3 months | baseline, 1 month, 3 months
  Power Doppler assessment of selected synovial sites is carried out with settings standardized to a pulse repetition frequency of 700 Hz. The intensity of the blood flow in the synovium is scored into 0 to 3 (0=No flag; 1 = 1 flag; 2 = 2-3 flags; 3=>3 flags) adapted from Klukowska and Melchiorre et al
Short Form -36 score and Change from Baseline at 1 & 3 months | baseline, 1 month, 3 months
  The SF-36 is filled out taking into account the person's condition in the last one month and scores range from 0 to 100, with higher scores indicating better health-related quality of life.
Hemophilia Joint Health Score (HJHS) and Change from Baseline at 1 & 3 months | baseline, 1 month, 3 months
  The HJHS is a structured physical examination score evaluating the joint health in hemophilia patient. The score for each joint is the sum of the individual items including swelling, swelling duration, muscle atrophy, axial alignment, crepitus of motion, flexion loss & extension loss, joint pain and strength. A score of 20 suggests the worst possible damage/impairment in the evaluating joint.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Ying Li, Principal Investigator — Hemophilia care and research center
Locations (1):
- Hemophilia care and research center, Taipei, Taiwan